CLINICAL TRIAL: NCT04974021
Title: An Open Label,Single-center, Non-interventional Prospective Study to Determine the Efficacy of Iron Therapy Using Intravenous Ferric Carboxymaltose and Its Effect in Reducing Arrhythmic Events in Participants With Iron Deficiency and HFrEF
Brief Title: Iron Intravenous Therapy in Reducing the Burden of Severe Arrhythmias in Heart Failure With Reduced Ejection Fraction
Acronym: RESAFE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Other Study IDs: 219/12-3-19
Record Dates: First submitted 2021-07-05; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Ferric Carboxymaltose; Heart Failure With Reduced Ejection Fraction; Arrhythmias, Cardiac
Keywords: ferric carboxymaltose; heart failure; arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Failure | interventions — ferric carboxymaltose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants: HFrEF patients undergoing iron therapy with intravenous carboxymaltose (FCM). FCM administered dosage as per clinical routine. FCM administration is repeated no sooner than 3 months than last therapy, based on repeat ferritin and transferrin saturation levels.
  Interventions: Drug: Ferric carboxymaltose

INTERVENTIONS:
Drug: Ferric carboxymaltose — Intravenous ferric carboxymaltose for the treatment of iron deficiency in HFrEF as per 2016 European Society of Cardiology Heart Failure guidelines.
  Other Names: Ferinject

SUMMARY:
An open label,single-center, non-interventional prospective study with the aim on investigating the effect of intravenous ferric carboxymaltose in restoring iron status and reducing the risk of severe arrhythmic events in participants with iron deficiency and a reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
Patients with HFrEF already scheduled to receive IV FCM to treat iron deficiency will be included in this registry trial. These patients undergo clinical examination, echocardiography, blood testing, 6-minute walking testing, cardiopulmonary exercise testing, cardiac implantable device interrogation, 24-hour Holter monitoring and quality of life quantification as part of standard clinical practice. This database will be extracted from clinical databases and stored on a separate, registry database. The study will examine the effect of IV FCM on patients' iron stores, arrhythmic burden, hospitalizations and clinical, echocardiographic, exercise-testing-derived and biological markers of disease severity such as 6-minute walking distance, peak VO2 consumption, LVEF and LV global longitudinal strain and NT-proBNP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HFrEF (LVEF≤40%)
* Implanted cardiac implantable electronic device with at least 3 months of recorded arrhythmic history
* Patient is scheduled to receive IV ferric carboxymaltose to treat diagnosed iron deficiency

Exclusion Criteria:

* Myocardial infarction, acute heart failure or life-threatening arrhythmias in the preceding 15 days
* Autoimmune disorders, cancer or other diseases other than heart failure that significantly affect patients' life expectancy, appetite and emotional status
* Known allergic reaction to ferric carboxymaltose.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure and reduced ejection fraction, cardiac implantable electronic devices and iron deficiency visiting the outpatient HF clinic of the Third Department of Cardiology AUTh
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | 6 and 12 months
  Measured in g/dL, will be aggregated to form a composite primary endpoint of hemoglobin ≥ 12g/dL, plasma ferritin ≥ 50 ng/mL and transferrin saturation > 20%
Ferritin | 6 and 12 months
  Measured in ng/mL, will be aggregated to form a composite primary endpoint of hemoglobin ≥ 12g/dL, plasma ferritin ≥ 50 ng/mL and transferrin saturation > 20%
Transferrin saturation | 6 and 12 months
  Measured as a percentage, will be aggregated to form a composite primary endpoint of hemoglobin ≥ 12g/dL, plasma ferritin ≥ 50 ng/mL and transferrin saturation > 20%

SECONDARY OUTCOMES:
HF-related hospitalizations | 6 and 12 months
  Hospitalizations due to acute-on-chronic heart failure or worsening heart failure (compared with 12 months preceding treatment)
N-terminal prohormone of brain natriuretic peptide (NT-proBNP) | 6 and 12 months
  NT-proBNP levels measured in serum (compared to baseline). NT-proBNP values are reported in pg/mL.
Kansas City Cardiomyopathy Questionnaire | 6 and 12 months
  HF-specific QoL quantified with the Kansas City Cardiomyopathy Questionnaire (compared to baseline). The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status. The questionnaire ranges from 0% (worst possible QoL) to 100% (best possible QoL)
EQ-5D-5L | 6 and 12 months
  General QoL is quantified with the EQ-5D-5L questionnaire (compared to baseline). EQ-5D-5L is a standardised measure of health-related quality of life. It contains a short descriptive system questionnaire and a visual analogue scale (EQ VAS). VAS ranges 0% to 100%.
Ventricular tachycardias recorded by cardiac implantable electronic device | 6 and 12 months
  Compared with 12 months preceding recruitment.
Non-sustained ventricular tachycardias recorded by cardiac implantable electronic device | 6 and 12 months
  Compared with 12 months preceding recruitment.
Appropriate therapies administered by cardiac implantable electronic device | 6 and 12 months
  Compared with 12 months preceding recruitment.
Appropriate atrial mode switch events recorded by cardiac implantable electronic device | 6 and 12 months
  Compared with 12 months preceding recruitment.
Non-sustained ventricular tachycardias recorded during 24-hour Holter monitoring | 6 and 12 months
  Compared with baseline.
Ventricular runs recorded during 24-hour Holter monitoring | 6 and 12 months
  Compared with baseline.
Ventricular triple premature complexes during 24-hour Holter monitoring | 6 and 12 months
  Compared with baseline.
Ventricular dual premature complexes during 24-hour Holter monitoring | 6 and 12 months
  Compared with baseline.
Ventricular premature complexes during 24-hour Holter monitoring | 6 and 12 months
  Compared with baseline.
Left ventricular end-diastolic volume index (LVEDVi) | 6 and 12 months
  Compared to baseline. Measured in mL/m^2.
Left ventricular ejection fraction (LVEF) | 6 and 12 months
  Compared to baseline. Measured as a percentage.
Left ventricular mass index (LVMi) | 6 and 12 months
  Compared to baseline. Measured in g/m^2.
Left ventricular global longitudinal strain (LV GLS) | 6 and 12 months
  Compared to baseline. Measured as a percentage.
Peak early diastolic tissue velocity (e') | 6 and 12 months
  Μeasured at the septal and lateral mitral annulus. Used to calculate E/e' ratio. Measured as m/s.
E-wave mitral inflow velocity (E) | 6 and 12 months
  Used to calculate E/e' ratio. Measured as m/s.
Right ventricular fractional area change (RV FAC) | 6 and 12 months
  Compared to baseline. Measured as a percentage.
6-minute walking distance (6MWD) | 6 and 12 months
  Distance recorded during six-minute walk testing. Measured in meters. Compared to baseline.
Maximal oxygen consumption (VO2 max) | 6 and 12 months
  Maximal oxygen consumption recorded during cardiopulmonary exercise testing. Measured in mL/kg/min. Compared to baseline.
Minute ventilation/carbon dioxide production slope (VE/VCO2 slope) | 6 and 12 months
  The VE/VCO2 slope recorded during cardiopulmonary exercise testing. Absolute unit. Compared to baseline.
End-tidal carbon dioxide at anaerobic threshold (etCO2-AT) | 6 and 12 months
  Recorded during cardiopulmonary exercise testing. Measured in mmHg. Compared to baseline.
Late potentials | 6 and 12 months
  Signal Averaged ECG (SAECG) enables the detection of late potentials. Specialist software automatically performs the detection of late potentials in patients' Holter monitor recordings.
Microvolt T-wave Alternans (TWA) | 6 and 12 months
  Specialist software quantifies microvolt TWA voltage in patients' Holter monitor recordings. microvolt TWA is measured in μV.
Heart rate turbulence (HRT) | 6 and 12 months
  Heart rate turbulence (HRT) is the baroreflex-mediated short-term oscillation of cardiac cycle lengths after spontaneous ventricular premature complexes. Specialist software detects abnormal HRT in patients' Holter monitor recordings. The existence of abnormal heart rate turbulence is a nominal variable.
Deceleration capacity | 6 and 12 months
  (Heart rate) deceleration capacity is a measurement of autonomic nerve regulation in heart failure. Specialist software quantifies deceleration capacity, which is measured in milliseconds (ms).

CONTACTS AND LOCATIONS:
Overall Officials: Vassilios P Vassilikos, PhD, Principal Investigator — Hippokration General Hospital of Thessaloniki, Third Department of Cardiology, AUThi
Locations (1):
- Hippokration General Hospital of Thessaloniki, Third Department of Cardiology (Aristotle University of Thessaloniki), Thessaloniki, Macedonia, Greece

IPD SHARING:
Plan to Share IPD: Undecided